CLINICAL TRIAL: NCT03854396
Title: A Randomized, Double-blind, Placebo-controlled Trial on the Preventive Effect of Intravaginal Prasterone (DHEA, Intrarosa®) on Recurrent Urinary Tract Infections in Women With Genitourinary Syndrome of Menopause
Brief Title: Clinical Trial on the Preventive Effect of Intravaginal Prasterone on Recurrent Urinary Tract Infections in Postmenopausal Women
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: due to termination of ISR by PI with agreement by grant sponsor
Sponsor: Olivia Cardenas-Trowers, M.D. (Other)
Collaborators: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Olivia Cardenas-Trowers, M.D., Fellow Physician in Female Pelvic Medicine & Reconstructive Surgery, University of Louisville
Organization: University of Louisville (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 19.0075
Record Dates: First submitted 2019-02-24; First posted 2019-02-26 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Recurrent Urinary Tract Infection; Postmenopause; Postmenopausal Syndrome; Postmenopausal Symptoms; Menopause
Keywords: recurrent urinary tract infection; genitourinary syndrome of menopause; prasterone
MeSH Terms: conditions — Urinary Tract Infections | interventions — Dehydroepiandrosterone; witepsol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intravaginal prasterone insert (Active Comparator): Nightly intravaginal prasterone insert for 24 weeks
  Interventions: Drug: Prasterone
- Intravaginal placebo insert (Witepsol H-15) (Placebo Comparator): Nightly intravaginal placebo insert (Witepsol H-15, a mix of synthetic triglycerides) for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prasterone — Nightly intravaginal prasterone insert (6.5 mg prasterone at a concentration of 0.50%) for 24 weeks.
  Other Names: Intrarosa; Dehydroepiandrosterone; DHEA
  Arms: Intravaginal prasterone insert
Drug: Placebo — Nightly intravaginal placebo insert (Witepsol H-15, a mix of synthetic triglycerides) for 24 weeks.
  Other Names: Witepsol H-15; Witepsol
  Arms: Intravaginal placebo insert (Witepsol H-15)

SUMMARY:
Urinary tract infections (UTIs) are bothersome and more likely to occur in postmenopausal women. Frequent UTIs, as well as other problems with the urinary and genital systems such as painful sex and urinary frequency/urgency, are part of a symptom complex called genitourinary syndrome of menopause (GSM). Prasterone (Intrarosa®) is a man-made steroid that helps with painful sex in postmenopausal women. Because previous studies have shown prasterone to help with other GSM problems, this study was designed to investigate if prasterone used in the vagina decreases the number of UTIs in postmenopausal women.

DETAILED DESCRIPTION:
Urinary tract infections (UTIs) are costly contributing to more than 8 million ambulatory visits (84% women) in the United States in 2007. Recurrent urinary tract infections (rUTIs) are UTIs diagnosed on at least 2 urine cultures in 6 months, or at least 3 in 1 year. The incidence of rUTIs increases in menopause with an estimated 10-15% of women > 60 years old having rUTIs. rUTIs contribute to a constellation of bothersome genitourinary symptoms in some postmenopausal women called genitourinary syndrome of menopause (GSM). Thus, menopause, rUTIs, and GSM are intimately linked.

Prasterone (Intrarosa®) is a synthetic version of the steroid, dehydroepiandrosterone (DHEA), approved by the US Food and Drug Administration in 2016 for the treatment of moderate to severe dyspareunia due to GSM. Large, prospective studies have shown prasterone to safely decrease vaginal pH, decrease parabasal cells, increase superficial cells, and decrease symptoms related to atrophy like dyspareunia in women with GSM. Given prasterone's favorable treatment effects on some GSM symptoms, investigation of prasterone as a possible treatment option for rUTIs in the setting of GSM is warranted.

This is a single center, double-blind, placebo-controlled, randomized trial comparing the efficacy of nightly intravaginal prasterone for 24 weeks to intravaginal placebo in decreasing rUTIs in women with GSM. The study hypothesis is that intravaginal prasterone decreases UTI incidence in women with GSM compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older who are ≥ 1 year after spontaneous or surgical (bilateral oophorectomy) menopause
* Presence of ≤ 5% of superficial cells on vaginal smear and vaginal pH > 5.0
* History of ≥ 2 UTIs in 6 months or ≥ 3 UTIs in 12 months (with documentation of a UTI confirmed on urine culture within the past 1 year)
* Negative urine culture prior to treatment randomization

Exclusion Criteria:

* Known allergy/hypersensitivity to prasterone or its constituents
* Contraindications to estrogen: acute thrombophlebitis, history of blood clotting disorder, and/or personal history of thromboembolic disorder associated with estrogen use
* Known or suspected estrogen-dependent neoplasms or mammary, ovarian, cervical, or vaginal malignancies
* Known congenital urologic or gynecologic abnormality
* Chronic immunosuppression
* Need for chronic catheterization
* Vaginal bleeding of origin other than vaginal mucosal atrophy
* Vaginal infection requiring treatment
* Use of systemic hormone replacement therapy or estrogen within past 6 months
* Use of topical estrogen within past 3 months
* Consistent use of vaginal products (lubricants, douches)
* Ongoing antibiotic treatment
* Ongoing treatment with Lactobacillus
* Inability to comply with protocol or place vaginal insert with applicator appropriately
* Less than 3 months status post urinary incontinence and/or pelvic organ prolapse surgery
* Unable to speak or read English
* If an exclusion condition is resolved, the patient may be re-approached later for study recruitment (ie., genitourinary infection, use of antibiotics, etc)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of urinary tract infections (UTIs) | 12 weeks
  Rate of UTIs during the study with UTI defined as at least one symptom of UTI (eg., dysuria, urinary frequency/urgency/incontinence, hematuria) and at least ≥10^2 colony-forming units (CFUs)/mL of 1 or more uropathogens on urine culture.
Incidence of urinary tract infections (UTIs) | 24 weeks
  Rate of UTIs during the study with UTI defined as at least one symptom of UTI (eg., dysuria, urinary frequency/urgency/incontinence, hematuria) and at least ≥10^2 colony-forming units (CFUs)/mL of 1 or more uropathogens on urine culture.

SECONDARY OUTCOMES:
Mean days of antibiotic use | 12 weeks and 24 weeks
  Average number of days of antibiotic use for participants in each treatment group who develop a UTI.

OTHER OUTCOMES:
Change from baseline in treatment response as measured by the vaginal pH | Baseline, 12 weeks, and 24 weeks
  pH test strip.
Change from baseline in treatment response as measured by the percentage of parabasal cells in the maturation index of the vaginal smear | Baseline, 12 weeks, and 24 weeks
  Histological laboratory evaluation.
Change from baseline in treatment response as measured by the percentage of superficial cells in the maturation index of the vaginal smear | Baseline, 12 weeks, and 24 weeks
  Histological laboratory evaluation.
Change from baseline in treatment response as measured by the percentage of intermediate cells in the maturation index of the vaginal smear | Baseline, 12 weeks, and 24 weeks
  Histological laboratory evaluation.
Change from baseline in treatment response as measured by the Vulvovaginal Symptom Questionnaire (VSQ) | Baseline, 12 weeks, and 24 weeks
  21 items with four scales: symptoms, emotions, life impact, and sexual impact. Total scores range: 0-21 (higher scores suggestive of greater severity of symptoms).
Change from baseline in treatment response as measured by the self-reported most bothersome symptom (MBS) | Baseline, 12 weeks, and 24 weeks
  Via a questionnaire, patient rates symptoms of GSM that she experiences. The highest ranked symptom is the patient's MBS.
Change from baseline in treatment response as measured by the Overactive bladder questionnaire (OAB-q) | Baseline, 12 weeks, and 24 weeks
  Total scores range: 0-100 (higher scores on the symptom-severity scale suggestive of greater severity of symptoms and higher scores on the quality-of-life scale suggestive of better quality of life).
Change from baseline in treatment response as measured by the International Consultation on Incontinence Questionnaire-Urinary Incontinence-Short Form (ICIQ-UI-SF) | Baseline, 12 weeks, and 24 weeks
  Three items on frequency, amount of leakage, and overall impact. Scoring 0-21, higher values indicating increasing severity.
Number of participants with at least one adverse event | 12 weeks and 24 weeks
  Adverse events will only be those determined to be related to the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Cardenas-Trowers, M.D., Principal Investigator — University of Louisville; Sean L. Francis, M.D., Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Urogynecology at Springs Medical Center, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified raw data and other supporting materials will be made available to approved investigators. Email requests to olivia.cardenas-trowers@louisville.edu.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available beginning 1 month and ending 24 months following article publication.
Access Criteria: Available to investigators whose proposed use of the data is for individual participant data meta-analysis and has been approved by an independent review committee for this purpose. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Foxman B. Urinary tract infection syndromes: occurrence, recurrence, bacteriology, risk factors, and disease burden. Infect Dis Clin North Am. 2014 Mar;28(1):1-13. doi: 10.1016/j.idc.2013.09.003. Epub 2013 Dec 8. PMID 24484571
- [Background] Brubaker L, Carberry C, Nardos R, Carter-Brooks C, Lowder JL. American Urogynecologic Society Best-Practice Statement: Recurrent Urinary Tract Infection in Adult Women. Female Pelvic Med Reconstr Surg. 2018 Sep/Oct;24(5):321-335. doi: 10.1097/SPV.0000000000000550. No abstract available. PMID 29369839
- [Background] Iosif CS, Bekassy Z. Prevalence of genito-urinary symptoms in the late menopause. Acta Obstet Gynecol Scand. 1984;63(3):257-60. doi: 10.3109/00016348409155509. PMID 6730943
- [Background] Rahn DD, Carberry C, Sanses TV, Mamik MM, Ward RM, Meriwether KV, Olivera CK, Abed H, Balk EM, Murphy M; Society of Gynecologic Surgeons Systematic Review Group. Vaginal estrogen for genitourinary syndrome of menopause: a systematic review. Obstet Gynecol. 2014 Dec;124(6):1147-1156. doi: 10.1097/AOG.0000000000000526. PMID 25415166
- [Background] Portman DJ, Gass ML; Vulvovaginal Atrophy Terminology Consensus Conference Panel. Genitourinary syndrome of menopause: new terminology for vulvovaginal atrophy from the International Society for the Study of Women's Sexual Health and the North American Menopause Society. Menopause. 2014 Oct;21(10):1063-8. doi: 10.1097/GME.0000000000000329. PMID 25160739
- [Background] Portman DJ, Goldstein SR, Kagan R. Treatment of moderate to severe dyspareunia with intravaginal prasterone therapy: a review. Climacteric. 2019 Feb;22(1):65-72. doi: 10.1080/13697137.2018.1535583. Epub 2018 Dec 17. PMID 30554531
- [Background] Labrie F, Archer DF, Koltun W, Vachon A, Young D, Frenette L, Portman D, Montesino M, Cote I, Parent J, Lavoie L, Beauregard A, Martel C, Vaillancourt M, Balser J, Moyneur E; VVA Prasterone Research Group. Efficacy of intravaginal dehydroepiandrosterone (DHEA) on moderate to severe dyspareunia and vaginal dryness, symptoms of vulvovaginal atrophy, and of the genitourinary syndrome of menopause. Menopause. 2016 Mar;23(3):243-56. doi: 10.1097/GME.0000000000000571. PMID 26731686
- [Background] Labrie F, Martel C, Berube R, Cote I, Labrie C, Cusan L, Gomez JL. Intravaginal prasterone (DHEA) provides local action without clinically significant changes in serum concentrations of estrogens or androgens. J Steroid Biochem Mol Biol. 2013 Nov;138:359-67. doi: 10.1016/j.jsbmb.2013.08.002. Epub 2013 Aug 14. PMID 23954500
- [Background] Labrie F, Archer DF, Bouchard C, Girard G, Ayotte N, Gallagher JC, Cusan L, Baron M, Blouin F, Waldbaum AS, Koltun W, Portman DJ, Cote I, Lavoie L, Beauregard A, Labrie C, Martel C, Balser J, Moyneur E; Members of the VVA Prasterone Group. Prasterone has parallel beneficial effects on the main symptoms of vulvovaginal atrophy: 52-week open-label study. Maturitas. 2015 May;81(1):46-56. doi: 10.1016/j.maturitas.2015.02.005. Epub 2015 Feb 16. PMID 25771041